CLINICAL TRIAL: NCT05366959
Title: The Relationship Between Trunk Muscle Endurance and Physical Activity, Low Back Pain and Fatigue in Young Adults
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: 4
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Trunk muscle endurance; Low back pain; Fatigue; Physical Activity
MeSH Terms: conditions — Low Back Pain; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trunk Muscle Endurance test — Trunk flexors endurance test: Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated and the time it maintains this position will be recorded in seconds.
  Modified "Biering-Sorensen" test: With this test, the endurance of trunk extensors is evaluated. The subjects are positioned in the prone position with the pelvis, hips and knees on the bed. The subjects are asked to extend their upper body straight forward from the edge of the table and the time they maintain this position will be recorded in seconds.
  Lateral bridge test: During the test, the subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position, and the time they held the position would be recorded in seconds. The test will be done on both sides.
Other: Fatigue Severity Scale — "Fatigue Severity Scale" was used to evaluate the fatigue level of the participants. This scale consists of a 7-point Likert scale. 1 point means strongly disagree, 7 means strongly agree. High scores are associated with increased fatigue. Evaluates the effects of fatigue on physical function, motivation, family and social life. Turkish validity and reliability was established.
Other: Roland Moris Scale — The "Roland Moris Scale" will be used to evaluate the participants for low back pain assessment. The Roland Morris Inquiry Form was designed to evaluate the functional disability of the patient. The total score ranges from 0 (no disability) to 24 (severe disability). The higher the total score, the lower the patient's functionality. It is a questionnaire filled by the patient, which evaluates the functionality of 24 items questioning the patient's mobility, self-care and sleep status. Each item marked as 'Yes' is given 1 point, and answers marked as 'No' are given 0 points. Turkish validity and reliability was established.
Other: Physical Activity Levels — The physical activity level of the participants will be measured with the International Physical activity scale: MET values will be calculated according to this scale, which has Turkish validity and reliability.

SUMMARY:
The trunk is a kinetic link that facilitates the transmission of force and angular moments between the lower and upper extremities, provides proximal stability for distal mobility, and maintains balance by keeping the body weight within the support surface.While trunk muscle strength is important for maintaining daily living activities, trunk muscle endurance plays an important role in preventing injuries by stabilizing the spine during long-term physical activity and sports activities (2).Decreased trunk muscle endurance can result in fatigue and low back pain. Low back pain is a major public health problem worldwide. In modern industrial society, the number of low back pain patients is increasing due to sedentary lifestyles, lack of exercise and working conditions.The lifetime prevalence of low back pain has been reported as 84%.80% of low back pain is nonspecific, that is, muscle weakness and ligament-related reasons for unknown reasons(3,4).Increasing the endurance of the waist muscles with exercise is used in the treatment of low back pain. From this point of view, while planning our study, we wanted to evaluate whether the decrease in trunk muscles is associated with low back pain and fatigue in young adults.

DETAILED DESCRIPTION:
Our research will be carried out in healthy youngs adult volunteers between the ages of 18-24.It is a non-invasive cross-sectional observational study without a control group.

No device will be used.The following measurement and evaluation methods will be applied to all individuals who voluntarily agree to participate in the research.First, demographic data will be collected with the Patient Evaluation Form. For trunk endurance measurement, McGill Trunk Muscle Endurance Tests, Modified Biering-Sorensen test and Lateral bridge test will be used.These tests measure muscle strength in seconds with examination as described below and do not require a device.Fatigue severity scale and Roland Morris Disability Form will be filled to evaluate fatigue and lumbar network.Physical Activity level will be measured with the International Physical Activity Scale.

ELIGIBILITY:
Inclusion Criteria:

-Voluntarily agree to participate in the research

Exclusion Criteria:

* History of musculoskeletal surgery in the last 1 year
* Diagnosis of lumbar disc herniation, spondylolisthesis, knee ligament and connective tissue damage
* Scoliosis
* Pregnancy
* Malignancy and inflammatory disease

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our research is a cross-sectional study conducted on 201 healthy young adult university student volunteers aged 18-24.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Trunc Muscle endurance -Trunk flexors endurance test | 0 (baseline)
  Trunk flexors endurance test: Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated and the time it maintains this position will be recorded in seconds.
Trunc Muscle endurance -Modified "Biering-Sorensen" test: | 0 (baseline)
  Modified "Biering-Sorensen" test: With this test, the endurance of trunk extensors is evaluated. The subjects are positioned in the prone position with the pelvis, hips and knees on the bed. The subjects are asked to extend their upper body straight forward from the edge of the table and the time they maintain this position will be recorded in seconds.
Trunc Muscle endurance -Lateral bridge test. | 0 (baseline)
  Lateral bridge test: During the test, the subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position, and the time they held the position would be recorded in seconds. The test will be done on both sides.
Roland Morris Scale | 0 (baseline)
  The "Roland Moris Scale" will be used to evaluate the participants for low back pain assessment. The Roland Morris Inquiry Form was designed to evaluate the functional disability of the patient. The total score ranges from 0 (no disability) to 24 (severe disability). The higher the total score, the lower the patient's functionality. It is a questionnaire filled by the patient, which evaluates the functionality of 24 items questioning the patient's mobility, self-care and sleep status. Each item marked as 'Yes' is given 1 point, and answers marked as 'No' are given 0 points. Turkish validity and reliability was established.
Fatigue Severity Scale | 0 (baseline)
  "Fatigue Severity Scale" was used to evaluate the fatigue level of the participants. This scale consists of a 7-point Likert scale. 1 point means strongly disagree, 7 means strongly agree. High scores are associated with increased fatigue. Evaluates the effects of fatigue on physical function, motivation, family and social life. Turkish validity and reliability was established.
physical activity level | 0 (baseline)
  The physical activity level of the participants will be measured with the International Physical activity scale: MET values will be calculated according to this scale, which has Turkish validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asisst Prof, Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kırşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] .Abaraogu UO, Ugwa WO. Selected anthropometrics, spinal posture, and trunk muscle endurance as correlated factors of static balance among adolescent and young adult males. Turk J Phys Med Rehab. 2016;1:9-15.
- [Background] Martinez-Romero MT, Ayala F, Aparicio-Sarmiento A, De Ste Croix M, Sainz De Baranda P. Reliability of five trunk flexion and extension endurance field-based tests in high school-aged adolescents: ISQUIOS programme. J Sports Sci. 2021 Aug;39(16):1860-1872. doi: 10.1080/02640414.2021.1903706. Epub 2021 Mar 28. PMID 33775212
- [Background] Koumantakis GA, Malkotsis A, Pappas S, Manetta M, Anastopoulos T, Kakouris A, Kiourtsidakis E. Lumbopelvic sagittal standing posture associations with anthropometry, physical activity levels and trunk muscle endurance in healthy adults. Hong Kong Physiother J. 2021 Dec;41(2):127-137. doi: 10.1142/S1013702521500128. Epub 2021 May 4. PMID 34177201
- [Background] Abdelraouf OR, Abdel-Aziem AA. THE RELATIONSHIP BETWEEN CORE ENDURANCE AND BACK DYSFUNCTION IN COLLEGIATE MALE ATHLETES WITH AND WITHOUT NONSPECIFIC LOW BACK PAIN. Int J Sports Phys Ther. 2016 Jun;11(3):337-44. PMID 27274419